CLINICAL TRIAL: NCT01311271
Title: Effects of the Quantity of Repetitive Transcranial Magnetic Stimulation on the Recovery of Upper Motor Function After Stroke: a Randomized Controlled Trial
Brief Title: Effects of the Quantity of Repetitive Transcranial Magnetic Stimulation(rTMS) on the Recovery After Stroke
Status: Terminated | Phase: Phase 2 / Phase 3 | Type: Interventional
Why Stopped: Only two subjects have been recruited from start of the study. We decided to start the study in this topic, after revising the study protocol.
Sponsor: Seoul National University Bundang Hospital (Other)
Collaborators: Asan Medical Center (Other); Gyeongsang National University Hospital (Other); Hanyang University (Other); Seoul National University Boramae Hospital (Other)
Responsible Party: Principal Investigator, Nam-Jong Paik, Professor, Seoul National University Bundang Hospital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: E-1011-056-003
Record Dates: First submitted 2011-03-04; First posted 2011-03-09 (Estimated); Last update posted 2015-05-19 (Estimated); Status verified 2015-05

CONDITIONS: Stroke; Hemiplegia
Keywords: Stroke; Cerebrovascular disease; hemiplegia; Transcranial magnetic stimulation; repetitive transcranial magnetic stimulation; rTMS; rehabilitation; Upper Extremity
MeSH Terms: conditions — Stroke; Hemiplegia; Cerebrovascular Disorders | interventions — Transcranial Magnetic Stimulation

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Sham rTMS-Sham rTMS (Sham Comparator): Sham rTMS for 2 weeks
  Interventions: Device: repetitive transcranial magnetic stimulation (rTMS)
- Sham rTMS-Real rTMS (Experimental): Sham rTMS in the first week and real rTMS in the second week
  Interventions: Device: repetitive transcranial magnetic stimulation (rTMS)
- Real rTMS-Real rTMS (Experimental): Real rTMS for 2 weeks
  Interventions: Device: repetitive transcranial magnetic stimulation (rTMS)

INTERVENTIONS:
Device: repetitive transcranial magnetic stimulation (rTMS) — 1 Hz frequency, 15 minutes, intensity of 90% resting motor threshold, with one session a day,
  * Real: unaffected M1 hotspot
  * Sham: coil perpendicular to scalp
  Other Names: TAMAS

SUMMARY:
The aim of this multicentric double blind study (randomized study) is to demonstrate the relationship between the amount of rTMS and the efficacy in the treatment of upper extremity motor deficits of stroke patients.

DETAILED DESCRIPTION:
Repetitive transcranial magnetic stimulation (rTMS) can modulate excitability of the brain via non-invasive methods. In that sense, rTMS has been used to treat a variety of symptoms of stroke during last two decades. Especially, improvement of upper extremity function has been proved by many studies. However, it remains uncertain about the optimum amount of rTMS.

The aim of this multicentric double blind study (randomized study) is to demonstrate the relationship between the amount of rTMS and the efficacy in the treatment of upper extremity motor deficits of stroke patients.

Fifty-seven patients will be included with written consent. After randomization, the subject will receive 3 different amount of treatment rTMS-rTMS, Sham-rTMS, Sham-Sham) in double blind methods.

ELIGIBILITY:
Inclusion Criteria:

* single mono-hemispheric ischemic or hemorrhagic stroke
* 1st onset stroke patient
* Upper extremity functional deficit attributable to acute stroke
* A stage of at least 3 on brunnström pre-treatment
* Written signed consent

Exclusion Criteria:

* Multiple lesion
* Bilateral cortical lesion and motor problems
* Cerebellar, or brainstem lesions
* History of more than one stroke
* Uncontrolled medical problems, such as: cardiopulmonary disease, severe rheumatoid arthritis, active joint deformity of arthritic origin, active cancer, or renal disease;
* Increased intracranial pressure
* History of seizure confirmed by interview and medical chart review
* Any individual who is on medication which is known to lower seizure threshold
* Other conditions that increase the risk of side effects due to rTMS procedures: a metal plate or metal object in the skull or eye, intracardiac line, increased intracranial pressure, cardiac pacemaker, implanted medication pump, tricyclic antidepressants, neuroleptics, history of seizure in the immediate family
* An age of less than 20 years old
* Any current actively treated medical or surgical condition or neurological or psychiatric illness other than stroke
* Complications that would prevent participation in the intervention, such as severe pain and severe spasticity
* Inability to cooperate outcome measure-related task
* Severe language disturbances
* Serious cognitive deficits
* Non-vascular cause for the neurological symptoms other central nervous system
* Disorder or peripheral neuropathy of the upper extremity
* Taking medication which interrupt brain activity
* Women who are pregnant

Ages: 20 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2 (Actual)
Dates: Start 2011-01; Primary Completion 2012-02 (Actual)

PRIMARY OUTCOMES:
Change in the Fugl-Meyer Assessment scale (upper extremity) | Baseline, weekly during treatment, at 4-week follow-up,and at 12-week follow-up

SECONDARY OUTCOMES:
Change in grip strength, lateral pinch force, tip pinch force, Purdue pegboard test, K-MBI, mRS,and brunnström stage | Baseline, weekly during treatment, at 4-week follow-up,and at 12-week follow-up

CONTACTS AND LOCATIONS:
Overall Officials: Nam-Jong Paik, MD, PhD, Principal Investigator — Seoul National University Bundang Hospital
Locations (1):
- Seoul National University Bundang Hospital, Seongnam-si, Gyeonggi-do, South Korea